CLINICAL TRIAL: NCT07247344
Title: Digital Phenotyping and Multimodal Biomarker Discovery for Major Depressive Episodes in Adolescent Inpatients: A Prospective Cohort Study
Brief Title: Multimodal Phenotyping in Adolescent Inpatient Depression: An Observational Study
Acronym: MAPS-IO
Status: Recruiting | Type: Observational
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Principal Investigator, Fei Wang, Professor, Jiangsu Province Nanjing Brain Hospital
Other Study IDs: 81725005-11
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-03

CONDITIONS: Adolescent; Major Depressive Disorder (MDD; Bipolar Disorder (BD)
Keywords: Major Depressive Episode
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: The diagnosis of Major Depressive Episode will be made according to the DSM-4 criteria. Neuroimaging assessment will be performed following standardized MRI quality control and interpretation procedures, jointly evaluated by an experienced radiologist and psychiatrist.
  Interventions: Other: data collection and follow-up

INTERVENTIONS:
Other: data collection and follow-up — Main measures and data collection methods:
  1. Recording of baseline demographic and clinical information of the participants.
  2. Multimodal magnetic resonance imaging.
  3. Heart rate variability.
  4. Electroencephalography.
  5. Emotion-related questionnaires.
  6. Cognitive tests.
  7. Behavioral data collection using wearable devices.
  8. Blood samples collection.

SUMMARY:
This cohort study involves the dynamic collection of clinical information from adolescent patients with major depressive episodes (including both major depressive disorder and bipolar disorder), encompassing serum parameters, physiological-behavioral signals, neuroimaging data, and neuropsychological scales. The study aims to summarize the comprehensive clinical characteristics of this population, identify new risk factors, and establish multivariate predictive models for treatment response, cognitive and emotional impairments. Furthermore, this research will thoroughly investigate the underlying neural mechanisms linking clinical manifestations and neuroimaging features in major depressive episodes.

DETAILED DESCRIPTION:
Research Objectives：

1. To conduct a longitudinal investigation in adolescent patients with major depressive episodes (including major depressive disorder and bipolar disorder) to observe the dynamic progression of cognitive function, emotional disorders, physiological-behavioral characteristics, and related contributing factors.
2. To systematically explore and summarize the clinical, physiological-behavioral, and neuroimaging characteristics of adolescents with major depressive episodes, with the aim of identifying novel risk factors associated with treatment response and clinical outcomes.
3. To perform an in-depth investigation into the underlying neurobiological mechanisms of major depressive episodes and examine the interrelationships between clinical manifestations, physiological-behavioral indicators, and neuroimaging outcomes.
4. To develop a multifactorial predictive model for treatment response and cognitive-emotional impairments in major depressive episodes, integrating clinical, physiological-behavioral, neuroimaging, and biomarker data.

ELIGIBILITY:
Inclusion Criteria:

* Between 10 and 20 years of age;
* Diagnosis of major depressive disorder (MDD) or bipolar disorder (BD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV). Diagnosis is assessed using the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I) for participants aged ≥18 years, or the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime version (K-SADS-PL) for participants aged <18 years;
* Current moderate to severe depressive episode, defined as Hamilton Depression Rating Scale (HAMD) score ≥17;
* Participants and 1 or 2 parents (patients' age< 18 years old) provide informed consent after the detailed description of the study.

Exclusion Criteria:

* Prior treatment with repetitive transcranial magnetic stimulation (rTMS), transcranial direct current stimulation (tDCS), electroconvulsive therapy (ECT), or standard psychological therapy within 6 months prior to screening;
* Comorbidity with other DSM-IV Axis I disorders or personality disorders;
* Judged clinically to be at serious risk of suicide;
* Diabetes mellitus, hypertension, vascular and infectious diseases and other major medical comorbidities;
* Unstable medical conditions, e.g., severe asthma; Neurological disorders, e.g., history of head injury with loss of consciousness for ≥ five minutes, cerebrovascular diseases, brain tumors and neurodegenerative diseases;
* Mental retardation or autism spectrum disorder;
* Contraindications to MRI (e.g., severe claustrophobia, pacemakers, metal implants);
* Current drug or alcohol abuse or dependence;
* Pregnant or lactating females.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will recruit participants aged 10-20 years diagnosed with major depressive disorder (MDD) or bipolar disorder (BD) according to DSM-IV criteria. Diagnoses will be confirmed using SCID-I (age ≥18) or K-SADS-PL (age <18).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
The 17-item Hamilton Depression Rating Scale (HAMD-17) | at baseline, week 1, week 2, week 4, week 24, and up to 1 year
  The HAMD-17 scale has 17 items. The total score ranges from 0-52, with higher score indicating more severe depressive symptoms. A total score of 0-7 is considered to be normal. Scores of 17 or higher indicate moderate, severe, or very severe depression.
Change in brain functional connectivity measured by resting-state functional MRI | at baseline, week 1, week 2, week 4, week 24, and up to 1 year
  Resting-state functional magnetic resonance imaging (rs-fMRI) will be employed to evaluate functional connectivity alterations in core brain networks
Change in Heart Rate Variability (HRV) via wearable device | Within 4 weeks, but not exceeding 1 year.
  Change in HRV derived from interbeat intervals (IBIs) collected via wearable device.
Change in daily step count and activity patterns recorded via wearable device | Within 4 weeks, but not exceeding 1 year.
  Change in daily step count and overall activity patterns automatically recorded via wearable device.
Change in Cytokines (reported in pg/mL) | at baseline, week 1, week 2, week 4, week 24, and up to 1 year
  Peripheral blood biomarkers will be measured to evaluate inflammatory and immune responses to treatment. Interferon-α (IFN-α) Interferon-γ (IFN-γ) Interleukin-1β (IL-1β) Interleukin-2 (IL-2) Interleukin-4 (IL-4) Interleukin-5 (IL-5) Interleukin-6 (IL-6) Interleukin-8 (IL-8) Interleukin-10 (IL-10) Interleukin-17 (IL-17) Tumor necrosis factor-alpha (TNF-α)
Change in Composite Immune-Inflammatory Ratio Index (unitless) | at baseline, week 1, week 2, week 4, week 24, and up to 1 year
  This composite index includes platelet-to-lymphocyte ratio (PLR), neutrophil-to-lymphocyte ratio (NLR), and monocyte-to-HDL cholesterol ratio (MHR), which together reflect systemic inflammatory activity and immune status.

SECONDARY OUTCOMES:
Change in electroencephalographic (EEG) activity measured by resting-state EEG | at baseline, week 1, week 2, week 4, week 24, and up to 1 year
  EEG recordings will be obtained before and after the treatment to evaluate changes in neural oscillatory activity and functional connectivity, including metrics such as power spectral density (alpha, beta bands), coherence, and event-related potentials.
Change from baseline in the Clinical Global Impression-Severity scale (CGI-S) | at baseline, week 1, week 2, week 4, week 24, and up to 1 year
  The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.
Change from baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) | at baseline, week 1, week 2, week 4, week 24, and up to 1 year
  MADRS is a clinician-rated scale used to assess depressive symptom severity and detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is rated from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms). The total score of MADRS ranges from 0 to 60, with higher score indicating more severe depression.
The Young Mania Rating Scale (YMRS) | at baseline, week 1, week 2, week 4, week 24, and up to 1 year.
  he Young Mania Rating Scale (YMRS) is an 11-item clinician-rated scale used to assess the severity of manic symptoms. Each item is scored from 0 to 4 or 0 to 8, depending on symptom intensity, with a total score ranging from 0 to 60. Higher scores indicate more severe manic symptoms. A score below 12 is generally considered to reflect remission or minimal symptoms.
Change in Blood Oxygen Saturation | Within 4 weeks, but not exceeding 1 year.
  Change in continuously monitored SpO₂ values from wearable sensors.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang, Study Chair — the Affiliated Nanjing Brain Hospital, Nanjing Medical University
Locations (1):
- 210000, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No